CLINICAL TRIAL: NCT04184193
Title: Benefits of Pulmonary Rehabilitation in Patients With Severe Lymphangioleiomyomatosis (LAM) - a Retrospective Analysis
Brief Title: Benefits of Pulmonary Rehabilitation in Patients With Severe Lymphangioleiomyomatosis (LAM)
Status: Completed | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr., Schön Klinik Berchtesgadener Land
Other Study IDs: LAM Trial
Record Dates: First submitted 2019-11-11; First posted 2019-12-03 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Lymphangioleiomyomatosis; LAM; Pulmonary Rehabilitation
MeSH Terms: conditions — Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Rehabilitation
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Patients will perform a comprehensive, inpatient pulmonary rehabilitation program for 4 weeks duration

SUMMARY:
Data from patients with the orphan disease of lymphangioleiomyomatosis (LAM) which performed a pulmonary Rehabilitation program will be analyzed retrospectively. Data will be taken from the internal data base of the reference Center (Schoen Klinik Berchtesgadener Land, Schoenau, Germany) where These data were collected during clinical routine. Data will be included from the year 2000 until now. A retrospectively matched COPD cohort will be included for comparison.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Lymphangioleiomyomatosis
* performed a pulmonary Rehabilitation program at the reference center

Exclusion Criteria:

* missing data
* repeated stay for pulmonary Rehabilitation at the reference center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a confirmed diagnosis of Lymphangioleiomyomatosis
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline 6 Minute walk distance at week 4 | baseline and week 4
  the walked distance in meter will be the Primary outcome of the 6 Minute walk test
Change from baseline Quality of life at week 4 | baseline and week 4
  the physical and mental health component summary score from the Short Form 36 Health Questionnaire will be recorded. Score range from 0 to 100 with lower scores indicating worse impairment

SECONDARY OUTCOMES:
Change from baseline lung function at week 4 | baseline and week 4
  forced expiratory volume in 1 second and inspiratory vital capacity will be provided in Liter and percent predicted

CONTACTS AND LOCATIONS:
Overall Officials: Rembert A Koczulla, MD, Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

REFERENCES:
- [Derived] Gloeckl R, Nell C, Schneeberger T, Jarosch I, Boensch M, Watz H, Wirtz H, Welte T, Kenn K, Koczulla AR. Benefits of pulmonary rehabilitation in patients with advanced lymphangioleiomyomatosis (LAM) compared with COPD - a retrospective analysis. Orphanet J Rare Dis. 2020 Sep 22;15(1):255. doi: 10.1186/s13023-020-01540-3. PMID 32962746